CLINICAL TRIAL: NCT07214038
Title: A Clinical Study to Evaluate the Stain Reduction Efficacy of a Non-Fluoride Tooth Whitening Dentifrice Containing Nano-Hydroxyapatite (nHAp) and a High Cleaning Silica Abrasive System Compared to a Commercial Fluoride Non-Whitening Dentifrice as a Negative Control
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boka LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GHRG-BOKA-STAIN-2025/01; GHRG-BOKA-STAIN-2025/01 (Other: Global Health Research Group H 8 Masjid Moth, GK-2, New Delhi, 110048, India)
Record Dates: First submitted 2025-09-24; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: Teeth Color; Teeth Staining
MeSH Terms: conditions — Tooth Discoloration | interventions — Toothpastes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Toothpaste (Experimental): Toothpaste with stain removing abilities. Toothpaste contains an abrasive system that provides increased stain removal capabilities. Product will be used by teh subject at home with a toothbrush. Instructions provided for daily use of the paste with the brush. Example brushing for two minutes per occasion.
  Interventions: Other: toothpaste
- Paste Dentifrice (Placebo Comparator): Toothpaste with No stain removing abilities. The abrasive system used in teh placebo, though having cleaning properties, will not have teh ability to remove excessive stain.
  Interventions: Other: toothpaste

INTERVENTIONS:
Other: toothpaste — toothpaste with stain removing abilities

SUMMARY:
To determine whether brushing with a non-fluoride tooth whitening dentifrice containing nHAP and a high cleaning silica system produces a greater level of stain reduction as indicated by the Modified Lobene Stain Index (MLSI) for the overall tooth surfaces than brushing with a commercial fluoride toothpaste for a period of 2 weeks.

DETAILED DESCRIPTION:
To determine whether brushing with a non-fluoride tooth whitening dentifrice containing nHAP and a high cleaning silica system produces a greater level of stain reduction as indicated by the Modified Lobene Stain Index (MLSI) for the overall tooth surfaces than brushing with a commercial fluoride toothpaste for a period of 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

Consent Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.

2) Age Aged at least 18 years.

3) Compliance Understands and is willing, able and likely to comply with all study procedures and restrictions.

4) General Health Good general health with no clinically significant and relevant abnormalities of medical history or dental examination in the opinion of the investigator or dental assessor.

5) Dental Details

1. Good oral health with 16 natural teeth including 11 of the 12 anterior teeth.
2. All facial surfaces gradable with no large restorations as judged by the investigator or dental assessor.

Exclusion Criteria:

Pregnancy Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.

2) Breast-feeding Women who are breast-feeding.

3) Allergy/Intolerance Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.

4) Clinical Study/Experimental Medication

1. Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit.
2. Previous participation in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
WHITENING | 2 WEEKS
  To determine whether brushing with a whitening dentifrice containing a high cleaning silica system produces a greater level of stain reduction as indicated by the Modified Lobene Stain Index (MLSI) Area x Intensity score for the overall tooth surfaces than brushing with a commercial fluoride non-whitening dentifrice as a negative control for 2 weeks.
TOOTH COLOR | 2 WEEKS
  TOOTH WHITENING AND ORAL OIFT TISSUE INTEGRITY
  To determine the oral soft tissue (OST) tolerance of the dentifrices.
  To compare the change from baseline in stain levels as represented by the MLSI scores for overall, gingival, interproximal and body areas of the facial and lingual surfaces for each dentifrice after 2 weeks of product use.

CONTACTS AND LOCATIONS:
Overall Officials: ASHISH KAKAR, BDS, Principal Investigator — GHRG
Locations (1):
- Global Health Research Group, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided